CLINICAL TRIAL: NCT00998218
Title: The Effect of Ranolazine on Cardiac Arrhythmias and Microvolt T- Wave Alternans in Patients With Significant Left Ventricular Dysfunction
Brief Title: Effect of Ranolazine on Arrhythmias and Microvolt T- Wave Alternans (MVTWA) Patients With LV Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aspirus Heart and Vascular Institute-Research and Education (Other)
Responsible Party: Principal Investigator, Karen Olson, Research Manager, Aspirus Heart and Vascular Institute-Research and Education
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAN-Twave alt
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Sudden Cardiac Death; Ventricular Arrythmias
Keywords: Sudden Cardiac Death; Arrythmias; Triggered activity; left ventricular dysfunction
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Dysfunction, Left | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Experimental): Ranolazine at 1000 mg BID (or 500 mg BID if the 1000 mg dose was not tolerated) for 4 weeks
  Interventions: Drug: Ranolazine
- Sugar pill (Placebo Comparator): Placebo comparator BID for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine at 1000 mg BID (or 500 mg BID if the 1000 mg dose was not tolerated) or a comparable placebo for the next 4 weeks
  Arms: Ranolazine
Drug: Placebo — Ranolazine at 1000 mg BID (or 500 mg BID if the 1000 mg dose was not tolerated) or a comparable placebo for the next 4 weeks
  Arms: Sugar pill

SUMMARY:
The purpose this investigation is to more thoroughly investigate the effects of ranolazine on arrhythmias and microvolt t-wave alternans in patients who have an automatic implantable cardioverter defibrillator (AICD) implanted either prophylactically to prevent sudden cardiac death, as well as in patients who may have had a clinically significant arrhythmic event prompting the insertion of the automatic implantable cardioverter defibrillator. It is anticipated this study will provide valuable new insight into the potential use of ranolazine to treat arrhythmias in higher risk patients.

DETAILED DESCRIPTION:
The device clinic of Aspirus Wausau Hospital follows approximately 2800 patients with pacemakers and automatic implantable cardioverter defibrillators (AICD). Approximately 300 of these patients have had an AICD inserted for primary or secondary arrhythmia prevention. From these 300 patients, approximately 20 patients who have an AICD implanted either prophylactically or for an established malignant arrhythmia will be recruited for this short study.

This is a study to investigate the effect of ranolazine on arrhythmias detected by their device to see if it will reduce abnormal beats. It will also study whether ranolazine will impact microvolt t-wave alternans (MVTWA), a measure of the tendency to have a serious arrhythmia. Approximately 10 patients with ischemic cardiomyopathy and 10 patients with a non-ischemic cardiomyopathy will be chosen. All will have an ejection fraction of 40% or less. Prior to institution of ranolazine, a MVTWA study will be performed (Cambridge Heart Inc.®). The AICD will be used to generate the increase in the heart rate needed to induce MVTWA. Each patient will have MVTWA assessed at 80 beats/minute and then again at 110 beats/minute. To eliminate interpretation bias, the auto interpretation feature of the MVTWA device will be used to determine whether the study is positive (MVTWA present) or negative (MVTWA absent) or indeterminate. In the coarse of this study, each patient will undergo a total of 3 MVTWA studies in an identical manner using the AICD to provide the needed changes in heart rate.

After informed consent is obtained the patient will begin a 10-day "ranolazine run in". Each randomized participant will be given a 10-day supply of ranolazine to make certain they tolerate the medication (constipation is by far the most common limiting side effect). Each participant will be started on 500 mg BID and after 3 days increased to 1000 mg BID. Participants able to tolerate at least 500 mg BID will then be considered eligible to participate in the study and randomly assigned to either ranolazine at 1000 mg BID (or 500 mg BID if the 1000 mg dose was not tolerated) or a comparable placebo for the next 4 weeks.

At least 3 days after the run in and prior to randomization, each patient will be brought in for or the baseline MVTWA and the device clinic will purge the AICD of data and reset the data counter. The patient will then immediately begin either placebo or ranolazine according to randomization. After 4 weeks, the MVTWA study will be repeated on either placebo or ranolazine and the arrhythmia data down loaded from the AICD, recorded and the arrhythmia counters and device operation counter again reset. Each patient will then cross over to the other therapy (ranolazine or placebo) for the next 4 weeks and the device interrogated and the MVTWA study repeated in an identical manner.

ELIGIBILITY:
Inclusion Criteria:

* Implant of AICD for the prevention of sudden cardiac death Implant of AICD for the prevention of sudden cardiac death

Exclusion Criteria:

* Any anti-arrhythmic agent (other than beta-blockers)
* History of or intolerance to ranolazine during the run in.
* History of severe constipation defined as requiring laxatives more than 5 times a week in order to have a bowel movement.
* Because of a weak inhibitory effect of ranolazine of the cytochrome p450, CYP 3A4, certain drugs metabolized by that system could accumulate. Although clinically significant interactions of ranolazine with these agents has not been demonstrated, patients on maximum doses of simvastatin, or patients on verapamil or diltiazem will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The effect of ranolazine compared to placebo on MVTWA and reproducibility of MVTWA will be demonstrated. A p value of < 0.05 will be considered significant | After 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: David K. Murdock, MD, Principal Investigator — Aspirus Heart and Vascular Institute-Research and Education
Locations (1):
- Aspirus Wausau Hospital, Wausau, Wisconsin, United States

REFERENCES:
- [Background] Tomaselli GF, Zipes DP. What causes sudden death in heart failure? Circ Res. 2004 Oct 15;95(8):754-63. doi: 10.1161/01.RES.0000145047.14691.db. PMID 15486322
- [Background] Ebinger MW, Krishnan S, Schuger CD. Mechanisms of ventricular arrhythmias in heart failure. Curr Heart Fail Rep. 2005 Sep;2(3):111-7. doi: 10.1007/s11897-005-0018-y. PMID 16138946
- [Background] Antzelevitch C, Belardinelli L, Zygmunt AC, Burashnikov A, Di Diego JM, Fish JM, Cordeiro JM, Thomas G. Electrophysiological effects of ranolazine, a novel antianginal agent with antiarrhythmic properties. Circulation. 2004 Aug 24;110(8):904-10. doi: 10.1161/01.CIR.0000139333.83620.5D. Epub 2004 Aug 9. PMID 15302796